CLINICAL TRIAL: NCT00056888
Title: Neurophysiological Studies in Patients With Psychogenic Movement Disorders
Brief Title: Neurophysiological Studies in Patients With Paroxysmal Hyperkinetic Movement Disorders
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030134; 03-N-0134
Record Dates: First submitted 2003-03-26; First posted 2003-03-26 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-02-17

CONDITIONS: Movement Disorders
Keywords: Electroencephalogram; Functional (BOLD) MRI; Startle Reflex; Electromyogram; Psychogenic; Paroxysmal; Dyskinesia; Kinesiogenic; EEG; Movement-Related Potential; Movement Disorder; Paroxysmal Hyperkinetic Movement; Disorder; Paroxysmal Dyskinesia
MeSH Terms: conditions — Movement Disorders; Dyskinesias; Disease; Chorea

SUMMARY:
This study will use three neurophysiological tests (see below) to determine what areas of the brain are responsible for paroxysmal hyperkinetic movement disorders. Patients with these disorders have sudden, brief attacks of movement, similar to epileptic seizures, but without loss of consciousness.

Normal volunteers and patients with two subtypes of paroxysmal hyperkinetic movement disorder, paroxysmal dyskinesia and psychogenic variant, that can be induced by a specific trigger, such as a sudden movement or prolonged exercise, will be included in this study. Candidates must be 12 years of age or older. Women of childbearing potential will be screened with a pregnancy test.

Participants will undergo one or more of the procedures detailed below. Patients' test results will be compared with those of normal volunteers. Before each test, participants will provide a medical history and undergo a brief physical examination. During each procedure, the subject will have surface electromyography (EMG) to measure the electrical activity of muscles. For EMG, electrodes (metal discs) filled with a conductive gel are taped to the skin over the muscle to be evaluated.

Functional Magnetic Resonance Imaging (fMRI)

MRI uses a strong magnetic field, radio waves, and computer technology to provide detailed images of the brain. For this test, the subject lies in a narrow cylinder (the scanner), while pictures of the brain are taken. Earplugs are worn to muffle loud noises caused by electrical switching of radio frequency circuits used in the scanning process. For functional MRI (fMRI), the subject is asked to mimic a movement that occurs during an attack, such as stiffening the hand to make a fist or flexing and rotating the arm inward, to detect changes in the brain regions involved in the movement. During the procedure, involuntary movements and voluntary movements will be monitored by surface EMG and by video camera. The test will last about 1-1/2 hours.

Electroencephalography (EEG)

EEG measures the electrical activity of the brain (brain waves) with electrodes placed on the scalp. During the procedure, muscle activity will be recorded with EMG. The subject will first relax and then will be asked to mimic a movement attack. The test will last from 1-1/2 to 2 hours.

Startle Reflex

The subject will put on a headphone and hear loud noises in a random fashion. During the test, muscle activity will be recorded with EMG and with a video c...

DETAILED DESCRIPTION:
Objective: The primary objective of this study is to determine the brain regions responsible during attacks for psychogenic paroxysmal hyperkinetic movement disorders using functional magnetic resonance imaging (fMRI). The secondary objective is to determine the neurophysiology during attacks for the same subjects compared to normal controls using electroencephalography (EEG) and Startle Reflex.

Study population: Psychogenic paroxysmal hyperkinetic movement disorder patients and a control group of healthy volunteers.

Design:

fMRI: Anatomical MRI and fMRI sequences are performed to obtain blood-oxygenation level-dependent (BOLD) imaging of brain activation during (1) triggered or provoked involuntary hyperkinetic movements and voluntary imitated movements in subjects with psychogenic paroxysmal hyperkinetic movement disorders and (2) voluntary imitated movements and rest states in healthy volunteers.

EEG: EEG will be recorded for jerk-locked back-averaging analysis.

Startle Reflex: Electromyography (EMG) will be recorded during exposure to auditory stimuli.

Outcome measures:

fMRI: BOLD will be obtained using baseline correction.

EEG

Startle Reflex: The latency, mean amplitude, and habituation of EMG amplitude will be measured.

ELIGIBILITY:
* INCLUSION CRITERIA:

Psychogenic paroxysmal hyperkinetic movement patients:

A. Established diagnosis of psychogenic hyperkinetic movement disorders. The diagnosis will be established by the preliminary screening in the NINDS Movement Disorders Outpatient Clinic, based on review of medical record, history, clinical evaluation, and videotapes of an attack.

B. Patients with clear onset stereotyped and defined hyperkinetic attacks.

C. Patients only with paroxysmal attacks of hyperkinetic movements.

D. Age 8 or older.

E. A reproducible trigger of paroxysmal hyperkinetic attacks, such as sudden movement, startle or prolonged exercise, which will produce attacks at least with 50% consistency.

F. Patients whose attacks can be precipitated easily.

G. Patients with typical attack involving unilateral extremities.

H. Patients taking medication that may influence the central nervous system, such as phenytoin, phenobarbital, carbamazepine, clonazepam, and antidepressants (but not limited to these) will be asked to hold the medication prior to the study. A sufficient drug washout period will be established dependant upon the individual drug. Subjects may be admitted to the NIH if necessary. They will be asked to abstain from alcohol and caffeine 24 hours prior to the study as well.

Normal Subjects:

A. Normal volunteers ranging from 8 to 65 will be included. Normal volunteers would be recruited from people who are registered as HMCS Normal Volunteers. All subjects should have a valid Clinical Center Medical Record Number.

B. Alcohol abstention is required for all subjects for both fMRI and EEG for 24 hours before the study.

EXCLUSION CRITERIA:

Psychogenic paroxysmal hyperkinetic patients:

A. Age younger than 8 years old.

B. Patients with attacks that involve head and neck movements, axial movements, bilateral limb involvement, or violent attacks that typically make patients fall to the ground. With respect to children, violent attacks are defined as any attack that can potentially result in injury (hitting the head, falls, violent flailing, hitting furniture or walls)

C. Previous history of or MRI findings consistent with brain tumors, strokes, trauma or arterial venous malformations.

D. Contraindication to MRI such as having devices not compatible with MRI (pacemaker, an implanted medical pump, brain stimulators, etc.), metallic prostheses in their body (metal pins and rods, heart valves, cochlear implants, etc.), and history of working with metals in the past, since such persons may potentially have small metal fragments in the eye without being aware of it.

E. Any diagnosis of progressive neurological disorders other than psychogenic paroxysmal hyperkinetic movement disorder.

F. Any history of significant medical disorders requiring chronic treatment with other drugs that affects the CNS, which cannot be stopped.

G. Women who are pregnant or nursing. Female subjects of childbearing potential (including all girls after menarche) will have specific interview and a pregnancy test prior to the study (before each imaging procedure if required) to ensure that they are not pregnant or nursing.

H. Any subject who is not capable of giving an informed consent. This will be determined at the initial evaluation at NINDS clinic. Patients with Mini Mental Score less than 25 or significant psychiatric history will be further evaluated by detailed neuropsychiatric testing, or consultation with a psychiatrist.

Normal Volunteers:

A. Normal subjects younger than 8 years and older than 65 will be excluded.

B. Normal subjects with MRI findings consistent with organic brain lesions such as brain tumors, stroke, trauma or AVMs will be excluded.

C. Normal subjects with a history of significant medical disorders such as cancers, or requiring continuous treatment with drugs will be excluded.

D. Subjects with mental disorders will be excluded.

E. We will not scan pregnant women because safety of high magnetic field to fetus is not established. Therefore, we will administer a urine pregnancy test for any female subjects of childbearing potential 24 hours prior to functional MRI scan.

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 115
Dates: Start 2003-03-21; Study Completion 2009-02-17

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Amjad AM, Halliday DM, Rosenberg JR, Conway BA. An extended difference of coherence test for comparing and combining several independent coherence estimates: theory and application to the study of motor units and physiological tremor. J Neurosci Methods. 1997 Apr 25;73(1):69-79. doi: 10.1016/s0165-0270(96)02214-5. PMID 9130680
- [Background] Andres FG, Mima T, Schulman AE, Dichgans J, Hallett M, Gerloff C. Functional coupling of human cortical sensorimotor areas during bimanual skill acquisition. Brain. 1999 May;122 ( Pt 5):855-70. doi: 10.1093/brain/122.5.855. PMID 10355671
- [Background] Berardelli A, Rothwell JC, Hallett M, Thompson PD, Manfredi M, Marsden CD. The pathophysiology of primary dystonia. Brain. 1998 Jul;121 ( Pt 7):1195-212. doi: 10.1093/brain/121.7.1195. PMID 9679773